CLINICAL TRIAL: NCT05094882
Title: Anatomical Location and Metastasis Pattern of Intrapulmonary Lymph Nodes in Non-small Cell Lung Cancer: a Multi-center, Prospective Observational Clinical Trial
Brief Title: Anatomical Location and Metastasis Pattern of Intrapulmonary Lymph Nodes in NSCLC (ECTOP-1010)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director, Fudan University
Other Study IDs: ALMPILN
Record Dates: First submitted 2021-10-04; First posted 2021-10-26 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Carcinoma; Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Intrapulmonary Lymph Nodes; Anatomical Location; Metastasis Pattern
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- RUL: patients who recieved the resection of right upper lobe (RUL)
  Interventions: Procedure: pulmonary lobectomy
- RML: patients who recieved the resection of right middle lobe ()
  Interventions: Procedure: pulmonary lobectomy
- RLL: patients who recieved the resection of right lower lobe (RML)
  Interventions: Procedure: pulmonary lobectomy
- LUL: patients who recieved the resection of left upper lobe (LUL)
  Interventions: Procedure: pulmonary lobectomy
- LLL: patients who recieved the resection of left lower lobe (LLL)
  Interventions: Procedure: pulmonary lobectomy

INTERVENTIONS:
Procedure: pulmonary lobectomy — resection of lung lobe

SUMMARY:
This is a clinical trial from Eastern Cooperative Thoracic Oncology Project (ECTOP), numbered as ECTOP-1010. Anatomical Location and Metastasis Pattern of Intrapulmonary Lymph Nodes (Group 11-13) in Non-small Cell Lung Cancer: a Multi-center, Prospective observational Clinical Trial

DETAILED DESCRIPTION:
Patients would be evaluated whether meet the criteria as clinical stage T1 non-small Cell Lung Cancer. Then, he/she would receive lobectomy. Finally, the detailed anatomical location of group 11-13 would be recorded immediately after surgery and their metastasis pattern would be explored in the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative examination showed patients with clinical T1 peripheral non-small cell lung cancer (NSCLC);
2. The lesion is located in a single lung segment or between two adjacent lung segments;
3. Perform radical lobectomy;
4. The preoperative examination did not reveal unresectable lymph nodes;
5. Have not received any other tumor-related treatments (including chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc.) before surgery;
6. No malignant tumor history;
7. No contraindications to surgery (ECOG score 0-1 points);

Exclusion Criteria:

1. Pathology revealed patients with non-T1 stage non-small cell lung cancer (NSCLC);
2. Radical lobectomy is not performed;
3. Acception of any anti-tumor treatment before surgery (excluding Chinese medicine treatment);
4. Refused to enter the group or asked to leave the group.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with stage T1 peripheral non-small cell lung cancer (NSCLC) undergoing radical lobectomy
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
metastasis rate of group 11-13 LN | one month after surgery
  metastasis rate of intrapulmonary lymph nodes (group 11-13 LN) in non-small cell lung cancer

SECONDARY OUTCOMES:
detailed anatomical location | immediately after surgery
  number of group 11-13 intrapulmonary lymph nodes in Non-small cell lung cancer and their detailed anatomical location

CONTACTS AND LOCATIONS:
Overall Officials: Hong Hu, Principal Investigator — Fudan University Affiliated Shanghai Cancer Center
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Inform Consent Form, Clinical Study Report would be shared every 3 months after the study begin.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: every 3 months after the study begin.